CLINICAL TRIAL: NCT06069505
Title: Detection of Azole Resistance Inducing Mutations on DNA Extracted Directly From Serum or Plasma of Immunocompromised Patients With an Invasive Aspergillus Infection Azole Resistance PCR Optimalization-study
Acronym: ARPO
Status: Recruiting | Type: Observational
Sponsor: Bart Rijnders (Other)
Responsible Party: Sponsor-Investigator, Bart Rijnders, Clinical Professor in Infectious Diseases, Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Other Study IDs: NL62004.078.17; MEC-2017-391 (Other: METC Erasmus Medical Center)
Record Dates: First submitted 2023-10-02; First posted 2023-10-05 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Invasive Aspergillosis
Keywords: invasive aspergillosis; PCR

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 80 ml of blood will be stored to analyze DNA extraction for PCR on serum and on plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Aspergillus PCR — Aspergillus PCR will be performed on different volumes of serum and plasma of patients with hematological malignancies with suspicion for invasive fungal infection.

SUMMARY:
Invasive aspergillosis (IA) is the most common mould infection in immunocompromised patients with haematological disease. Voriconazole, a triazole, improves overall survival of patients with an IA and is the mainstay of therapy. Resistance of A. Fumigatus emerged as an important clinical problem and infections with azole resistant Aspergillus have a high mortality. Nowhere in the world, azole resistance is more prevalent than in the Netherlands. Rapid detection of resistance is key to improve the patient's outcome but fungal cultures take time and are often negative. The investigators aim to detect azole resistance associated mutations in fungal DNA extracted directly from serum or plasma to accelerate diagnosis and improve outcome of patients infected with azole resistant A. fumigatus.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Lung CT shows lesions that fulfil the EORTC/MSG radiological criteria of possible invasive fungal infection.
* A bronchoalveolar lavage is planned or has been performed <48hrs earlier

Exclusion Criteria:

- Patients unable or unwilling to provide consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 100 haematology patients with a radiologically suspected invasive pulmonary aspergillosis and undergoing a bronchoalveolar lavage. After the BAL diagnostic tests have become available, confirmation of the suspected infection is expected in 25 patients and therefore 25 evaluable patients will remain. The investigators decided that another 50 patients should be included because only 25% had an invasive fungal infection after interim analysis of the first 50 patients included.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Performance of two different PCR test | 1 week
  The sensitivity and specificity will be determined of the different PCR's tested including the commercially available AsperGenius (Pathonostics, Maastricht) and the in-house PCR. For this purpose a patients diagnosed with proven or probable IPA according to the EORTC/MSG definition will be used as the gold standard.
Performance of two different media for the PCR test | 1 week
  Extraction medium (serum versus plasma) and extraction volume (1, 3 or 10 ml) that results in best sensitivity and specificity will be determined
Determination of best PCR cycle threshold | 1 week
  Extraction medium (serum versus plasma) and extraction volume (1, 3 or 10 ml) that results in best sensitivity and specificity will be determined

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus Medical Center (EMC), Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided